CLINICAL TRIAL: NCT03808077
Title: A Randomized Controlled Trial to Compare the Effectiveness of Deep vs. Moderate Neuromuscular Blockade in Reducing Postoperative Pain and Intra-Abdominal Insufflation Pressure During Minimally Invasive Robotic Prostatectomy
Brief Title: The Effect of Deep Versus Moderate Muscle Relaxants in Men During and After Robotic Surgery for Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-408
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; robotic surgery; muscle relaxants; neuromuscular blockade; 18-408; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Prostatic Neoplasms; Muscle Hypotonia | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Interventional Group: Deep Neuromuscular Blockade (Experimental): The Deep NMB group (Intervention) will have rocuronium infusion titrated to deep paralysis defined as PTC of 1-2 (infusion start rate 0.025mg/kg/min or 1.5mg/kg/hr).
  Interventions: Drug: Rocuronium 1.5mg/kg/hr
- Control Group: Moderate Neuromuscular Blockade (Active Comparator): The Moderate NMB group (Control ) will have rocuronium infusion titrated to moderate paralysis defined as TOF of 1-2 (infusion start rate 0.005mg/kg/min or 0.3mg/kg/hr).
  Interventions: Drug: Rocuronium 0.3mg/kg/hr

INTERVENTIONS:
Drug: Rocuronium 0.3mg/kg/hr — The Moderate NMB group (Control ) will have rocuronium infusion titrated to moderate paralysis defined as TOF of 1-2 (infusion start rate 0.003 mg/kg/min or 0.18mg/kg/hr).
  Arms: Control Group: Moderate Neuromuscular Blockade
Drug: Rocuronium 1.5mg/kg/hr — The Deep NMB group (Intervention) will have rocuronium infusion titrated to deep paralysis defined as PTC of 1-2 (infusion start rate 0.006mg/kg/min or 0.35mg/kg/hr).
  Arms: Interventional Group: Deep Neuromuscular Blockade

SUMMARY:
The purpose of this study is to determine if there is a difference in intra-abdominal pressure which surgeons use during surgery and post-surgery pain in men who undergo robotic prostate surgery with deep neuromuscular blockade (NMB), compared with moderate NMB.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients under the age of 80
* American Society of Anesthesiologists Physical Status 1, 2, 3.
* Elective Robotic Prostatectomy
* Patient undergoing surgery at Josie Robertson Surgical Center

Exclusion Criteria:

* Age younger than 18
* Inability to provide informed consent
* Allergy to rocuronium, sugammadex, midazolam, propofol, fentanyl, lidocaine, mannitol (IV Acetaeminophen), IV Acetaminophen, Ketorolac, Morphine, Hydromorphone, Dexamethasone, Zofran, Benadryl, Compazine
* Neuromuscular disease
* Any patient with previous abdominal surgery less than or equal to 20 years prior to scheduled surgery date
* Patients with BMI>35
* Severe renal impairment (Creatinine clearance < 30 ml/min)
* Patient receiving Toremifene or any history of receiving Toremifene
* Chronic pain patients
* Patients receiving suboxone
* Patients receiving succinylcholine

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rieth, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Tanaka A, Cai T, Platten M, Tollinche LE, DeJoy SJ. Anesthetic Management and Neuromonitoring in a Patient with Very Long-Chain Acyl-Coenzyme A Dehydrogenase Deficiency Undergoing Scoliosis Surgery: A Case Report and Review of Literature. Case Rep Anesthesiol. 2024 Jan 8;2024:1050279. doi: 10.1155/2024/1050279. eCollection 2024. PMID 38229914
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional Group: Deep Neuromuscular Blockade | Control Group: Moderate Neuromuscular Blockade
Started | 72 | 67
Completed | 67 | 63
Not Completed | 5 | 4
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Equipment Issues | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Group: Deep Neuromuscular Blockade | Control Group: Moderate Neuromuscular Blockade | Total
Number analyzed (Participants) | 72 | 67 | 139
Age, Continuous [Median (Full Range); unit: years] | 63 [44 to 73] | 63 [43 to 73] | 63 [43 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 72 | 67 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 68 | 59 | 127
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 60 | 52 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 67 | 139

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Intra-Abdominal Pressure (IAP) When Performing Robotic Prostatectomy in Participants Under a Moderate vs Deep Neuromuscular Blockade Technique
Description: Measured by continuous Intra-abdominal Pressure monitor in mmHg.
Time Frame: 6 hours post operation
Measure: Mean (Inter-Quartile Range); unit: mmHg
Arm/Group | Interventional Group: Deep Neuromuscular Blockade | Control Group: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 72 | 67
mmHg | 10.50 [8.93 to 12.71] | 11.41 [9.88 to 12.90]

2. Primary Outcome: Difference in Levels of Postoperative Pain in Participants Under a Moderate vs Deep Neuromuscular Blockade Technique During Robotic Prostatectomy Using the Pain Numeric Pain Scale (NPS).
Description: Difference in levels of postoperative pain in participants under a moderate vs deep Neuromuscular Blockade technique during robotic prostatectomy using the pain numeric pain scale (NPS). The numeric pain scale (NPS) is a subjective measure which can be used in recovery rooms to assist in the assessment of pain. Individuals rate their pain on an eleven-point scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Time Frame: 6 hours post operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interventional Group: Deep Neuromuscular Blockade | Control Group: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 72 | 67
score on a scale | 3.25 [1.90 to 4.14] | 3.41 [2.14 to 4.94]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Interventional Group: Deep Neuromuscular Blockade | Control Group: Moderate Neuromuscular Blockade
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/67
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/67
Other Adverse Events (participants affected / at risk) | 0/72 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional Group: Deep Neuromuscular Blockade (N=72) | Control Group: Moderate Neuromuscular Blockade (N=67)
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03808077/Prot_SAP_000.pdf